CLINICAL TRIAL: NCT00764712
Title: Comparison of Three Protocols for Tight Glycemic Control in Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Blaha, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POINT-protocols; GAUK no. 44407
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Hyperglycemia
Keywords: Tight glycemia control; cardiac surgery patients
MeSH Terms: conditions — Hyperglycemia | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Matias protocol (Active Comparator): A protocol based on the absolute glucose value - Matias protocol (Matias)
  Interventions: Drug: insulin
- Bath protocol (Active Comparator): A protocol based on the relative glucose change - Bath protocol (Bath)
  Interventions: Drug: insulin
- eMPC (Active Comparator): a computer-based model predictive control algorithm with variable sampling rate (eMPC)
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: insulin — Insulin was was administered according to each protocol rules/suggestions into a central venous line as a continuous infusion (Bath and eMPC protocols) or as a combination of a continuous infusion and boluses (Matias protocol). A standard concentration of 50 IU of insulin in 50 ml of 0.9% NaCl was used. In all patients, infusion of 10% glucose solution was initiated upon admission to ICU with glucose dose of 2.5 g/kg of ideal body weight (height in centimetres minus 100) per hour and lasted for 18 hours, when normal oral food intake was started. In ventilated patients, the glucose infusion lasted for 48 hours, and then standard enteral nutrition was initiated.
  Other Names: Actrapid HM, Novo Nordisk, Baegsvard, Denmark

SUMMARY:
A randomized trial to compare three insulin-titration protocols for tight glycemic control in surgical ICU: an absolute glucose (Matias) protocol, a relative glucose change (Bath) protocol, and an enhanced model predictive control algorithm (eMPC)

DETAILED DESCRIPTION:
120 consecutive post-cardiac surgery patients randomized to the three protocols with a target glycemia range from 4.4 to 6.1 mmol/l. Intravenous insulin was administered continuously or in combination with insulin boluses (Matias protocol). Blood glucose was measured in 1-4 hour intervals as requested by protocols.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the postoperative ICU after elective cardiac surgery

Exclusion Criteria:

* insulin allergy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The effectiveness of different TGC management protocols | ICU stay

SECONDARY OUTCOMES:
The safety with respect to hypoglycemia | ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Jan Blaha, MD, Principal Investigator — Charles University, Czech Republic
Locations (1):
- University Hospital in Prague, Prague, Czechia

REFERENCES:
- [Result] Blaha J, Kopecky P, Kotulak T, Kunstyr J, Matias M, Rubes D, Dobias M, Romaniv S, Kubatova J, Porizka M et al: Blood glucose control in cardiac surgery patients: a comparative study of different insulin protocols. Journal of Cardiothoracic and Vascular Anesthesia 2008, 22(S3):S23.